CLINICAL TRIAL: NCT06955715
Title: Pasteurized Donor Human Milk for HIV-Exposed Infants: A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Kelsey Cochrane, Principal Investigator, University of Saskatchewan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 106702
Record Dates: First submitted 2025-04-15; First posted 2025-05-02 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-04

CONDITIONS: HIV; Pregnancy; Breastfeeding; Infant Feeding Practices
Keywords: Donor Human Milk; HIV-Exposed Infants; Pasteurized Donor Milk; Infant Nutrition; Feasibility Study; HIV and Infant Feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: This study uses a single-group design where HIV-exposed infants receive pasteurized donor human milk as a supplement to infant formula or to support exclusive breastfeeding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pasteurized Donor Human Milk (Experimental): Pasteurized donor human milk sourced from the Norther Star Mother's Milk Bank (Calgary, AB, Canada)
  Interventions: Other: Pasteurized Donor Human Milk

INTERVENTIONS:
Other: Pasteurized Donor Human Milk — This is a single arm study in which all participants will receive pasteurized donor human milk sourced from the Norther Star Mother's Milk Bank (Calgary, AB, Canada)

SUMMARY:
Pasteurized Donor Human Milk (PDHM) is recognized as providing vital immunological and nutritional benefits to vulnerable infants. Although PDHM is widely used in neonatal intensive care units (NICUs) to prevent infections (necrotizing enterocolitis) and improve infant health outcomes, its use for other populations, such as HIV-exposed infants, has been minimal.

Pasteurized donor human milk is included in the 2023 Canadian Paediatric Society clinical consensus as a potential way to provide HIV-exposed infants some of the immunological benefits of human milk in a safe manner, as opposed to exclusive formula feeding (which is currently considered the gold standard for HIV-exposed infants). These new consensus guidelines also include recommendations to support those who wish to breastfeed using a harm reduction approach (e.g., increased viral load monitoring by peds infectious diseases), given the low risk of transmission in those adhering to antiretroviral medications. However, mixed feeding (e.g., breastfeeding and provision of infant formula) is not recommended, due to the potential for micro abrasions in the gastrointestinal epithelium as a result of the protein size in infant formula (which is larger and more abrasive than in human milk), which may increase the risk of HIV transmission if the HIV virus is present in breastmilk. As such, donor milk also presents a possible solution to support those who choose to breastfeed, but who may require a temporary supplement for whatever reason (e.g., nipple cracks, mastitis, etc.), as donor milk is human milk, thus has the same size of proteins and does not pose the same risk as infant formula in damaging the epithelial layer in the gut.

Overall, major obstacles remain that prevent newborns outside of the NICU from regularly having access to donor human milk. These obstacles are illustrated by the high cost of donor milk, which is not covered by government programs, and the lack of information about the clinical benefits (for both those who choose to breastfeed or formula feed), acceptability of caregivers for this feeding option, and feasibility of providing donor human milk outside of a hospital setting.

The investigators aim to determine whether giving PDHM to infants exposed to HIV is a practical possibility and learn from caregivers about any challenges associated with this feeding option. The results of this study will guide future research and a potential provincial initiative to expand access to PDHM for this population.

DETAILED DESCRIPTION:
The investigators will recruit women living with HIV who recently gave birth (or caregivers of HIV-exposed infants) living in Saskatoon, SK, Canada, and surrounding areas who are being followed by the Saskatchewan Health Authority (SHA) Pediatric Infectious Diseases. Women/caregivers may be currently formula feeding or breastfeeding their infant. PDHM will be provided to participants for a period of ~6-8 weeks (starting at ~2 months postpartum) and will involve 4 home visits to deliver PDHM in intervals of ~2-3 weeks and track feeding habits, as described below.

Visit 1 (Baseline; ~2 months postpartum): Deliver frozen PDHM to participant homes. For those who are formula feeding, we will provide 25 x 120 mL bottles, and for those who are breastfeeding, we will provide 8 x 120 mL bottles. Those who are formula feeding will be instructed to provide ~1-2 bottles of PDHM daily as a top-up to infant formula. Those who are breastfeeding will be instructed to provide PDHM as needed, if a supplement to breastfeeding is required for any reason (as opposed to supplementing with infant formula, which is not recommended for those breastfeeding). Caregivers will log the amount of PDHM given daily, any challenges, and any signs of poor tolerance (e.g., fussiness, vomiting, diarrhea). A baseline questionnaire will be given to collect demographic characteristics about the caregiver and birth data. Infant weight will be measured using a portable infant scale to establish a baseline for growth tracking.

Visit 2 (2-3 weeks) and Visit 3 (4-6 weeks): Collect all empty bottles from previous visits and completed tracking documents. Deliver a new batch of PDHM (quantities as described above).

Visit 4 (6-8 weeks; ~4 months postpartum): Collect all remaining empty bottles and final tracking documents. Infant weight using a portable infant scale will be measured to assess growth over the study period.

Participants will also receive a weekly check-in (phone call) to discuss any questions and gather general updates/information on infant feeding practices.

The investigators will further collect infant health related data collected by SHA Peds Infectious Disease as part of routine appointments. This will include anthropometric measurements (e.g., weight, height, head circumference) and occurrences of illness or opportunistic infections from birth to 4 months.

Statistical Analysis: We will calculate the mean ± SD (or median, IQR) for the frequency of donor milk provision (# of donor milk feedings/day) and volume (donor milk mL/day) based tracking documents; empty bottle counts will be used as a secondary estimate. Events of poor tolerance (e.g., colic, fussiness, vomiting) will be summarized using absolute frequencies and percentages. Any open-ended comments re: challenges, tolerance, or general thoughts re: provision of donor milk, will be categorized to identify trends among study participants. Clinical pilot data will include infant growth (e.g., mean ± SD daily weight gain velocity, percentiles for length-for-age, weight-for-age, head circumference, and weight-for-length) and reported rates of illness or infections, based on Pediatric Infectious Disease records.

ELIGIBILITY:
Inclusion criteria

* ≥15 years of age
* Pregnant or recently gave birth and living with HIV or is the primary caregivers of an HIV-exposed infant
* Being followed by SHA Pediatric Infectious Disease
* Saskatchewan resident (living within ~150 km from the University of Saskatchewan)
* Have a household freezer
* Willing to participate

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of PDHM provision (#/day) | 8-12 week intervention period
  Frequency (# of PDHM feedings/day) of PDHM provided to infants as a top up to infant formula or while breastfeeding
Volume of PDHM provision (mL/day) | 8-12 week intervention period
  Volume (mL/day) of PDHM provided to infants as a top up to infant formula or while breastfeeding

SECONDARY OUTCOMES:
Events of infant intolerance (n, %) | 8-12 weeks
  Participant reported events of poor tolerance (including gas, vomiting, diarrhea, etc.) which occur while providing the intervention (PDHM)
Caregiver-related experiences and challenges | 8-12 weeks
  Open-ended comments from caregivers regarding any concerns with PDHM provision (such as storage, thawing, preparation, or infant tolerance).

OTHER OUTCOMES:
Infant growth (g/day) | 8-12 weeks
  Infant growth (g/d weight gain) from visit 1 to visit 4 (baseline to endline)
Frequency of illness or opportunistic infections (n, %) | 8-12 weeks
  Rates of illness or opportunistic infection throughout the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey M Cochrane, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada